CLINICAL TRIAL: NCT05292469
Title: A Cluster Randomized Trial to Evaluate Comprehensive Approach to Hypertension Management in Nepal
Brief Title: Comprehensive Approach to Hypertension Management in Nepal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Institute for Implementation Sciences and Health, Kathmandu, Nepal (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 399476
Record Dates: First submitted 2022-03-09; First posted 2022-03-23 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Hypertension
Keywords: Nepal; Monitoring
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Cluster randomized Trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): Routine hypertension care
- Intervention arm (Experimental): Comprehensive approach to hypertension management that includes BP audit and feedback by physician (nurse and doctor), and patient support to monitor BP, and home based patient care by community health workers to encourage self-monitoring of BP followed by tailored educational counselling on behavioral and lifestyle change in addition to routine care.
  Interventions: Behavioral: Comprehensive approach to hypertension management

INTERVENTIONS:
Behavioral: Comprehensive approach to hypertension management — Trained health workers will review blood pressure (BP) logs and provide treatment. The patients will receive a BP lowering informational package, BP monitoring device and log book and pill-box and medication table. The participants will receive monthly home visits (6 visits) to discuss hypertension and ways to manage it. They will be encouraged to identify problems and developing an action plan to solve them. The participants will be encouraged to set behavioral goals. The follow up visits will review the progress made in implementing action plan and goals set and updating them. Review BP logs and facilitate tailored discussion on topics based on problems faced by participants on barriers to medication adherence, physical activity, weight management or diet. The family members will be involved and be accountable in supporting the patients in achieving the action plans.
  Arms: Intervention arm

SUMMARY:
Hypertension is a global risk factor for cardiovascular diseases. Approximately 80% hypertension burden is in low-and-middle income countries. Hypertension can be managed with antihypertensive medication and following effective lifestyle interventions, however the control rate of hypertension among those on treatment is dismal. In Nepal, a quarter of adult population have hypertension of whom, 44% are unaware of their status, 33% are on treatment, and, only 12% are controlled. A comprehensive intervention strategy for hypertension management has shown promising results in high income countries. Therefore, it is of interest to understand its effectiveness, appropriateness and feasibility in the low income settings such as Nepal. The objective of the trial is to assess the impact on net change in mean systolic blood pressure measured between 7 to 8 months follow-up of a comprehensive intervention which provides personalized counselling on lifestyle modification and medication adherence together with support for regular monitoring of blood pressure at home, compared with a control arm where hypertensive patients have access to routine care only. The investigators are proposing a cluster randomized controlled trial conducted in government health facilities from Budhanilakantha, an urban municipality in the Bagmati Province of Nepal. Trial arms: 1) control (routine hypertension care); 2) Comprehensive approach to hypertension management that includes blood pressure (BP) audit and feedback by physician (nurse and doctor), and patient support to monitor BP, and home based patient care by community health workers to encourage self-monitoring of BP followed by tailored educational counselling on behavioral and lifestyle change. Eligible participants providing consent will be enrolled into the trial by a research assistant who will conduct interviews. Those from the intervention arm will receive the home visits for 6 months. Participants from both arms will provide follow up data in 7 to 8 months.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension patients (systolic blood pressure 140 mmHg or more and/or diastolic blood pressure 90 mmHg or more on at least two separate visits, or use of antihypertensive medication)
* Living in the area served by the participating health facilities

Exclusion Criteria:

* Pregnancy
* Not able or willing to give informed consent,
* Critically ill from depilating conditions such as dialysis, cancer, palliative care
* Not likely to continue living in the area served by the health facility during trial follow up period (8 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1252 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-08-29 (Actual)

PRIMARY OUTCOMES:
Mean systolic blood pressure (BP) (mmHg) | Measured at baseline and follow up between 7 to 8 months after baseline
  Net change in mean systolic BP from baseline to follow up

SECONDARY OUTCOMES:
Mean diastolic BP (mmHg) | Measured at baseline and follow up between 7 to 8 months after baseline
  Net change in mean diastolic BP from baseline to follow up
Proportion controlling BP (<140/90 mmHg) | Measured at baseline and follow up between 7 to 8 months after baseline
  Proportion of participants controlling BP (<140/90 mmHg) from baseline to follow up
Waist Circumference (cm) | Measured at baseline and follow up between 7 to 8 months after baseline
  The mean difference in waist circumference measured at baseline and follow up
Body weight (Kg) | Measured at baseline and follow up between 7 to 8 months after baseline
  The mean difference in weight measured at baseline and follow up
Diet low in cholesterol, high in fruits and vegetables | Reported at baseline and follow up between 7 to 8 months after baseline
  The proportion consuming diet low in cholesterol, high in fruits and vegetables in the last 24 hours self reported at baseline and follow up
Daily salt intake (<1 teaspoon per day) | Reported at baseline and follow up between 7 to 8 months after baseline
  The proportion consuming less than 1 teaspoon of salt per day self reported at baseline and follow up
Medication adherence | Self reported at baseline and follow up between 7 to 8 months after baseline
  The proportion adhering to prescribed medication in the past two weeks measured at baseline and follow up
Physical activity | Self reported at baseline and follow up between 7 to 8 months after baseline
  The proportion engaged in moderate physical activity (2.5 hours per week) measured at baseline and follow up
Hypertension Knowledge Score | Self reported at baseline and follow up between 7 to 8 months after baseline
  All together 21 hypertension knowledge statement with 12 true false responses and others with multiple responses to create a aggregate score on hypertension Knowledge
Perceived Social Support Scale | Self reported at baseline and follow up between 7 to 8 months after baseline
  Twelve statements on perceived social support with 7 point Likert scale will be used at baseline and endline
Maintaining BP logs | Self reported at follow up between 7 to 8 months after baseline
  Proportion of trial participants maintaining self BP measurement logs asked during follow up

CONTACTS AND LOCATIONS:
Overall Officials: Solveig Kirsti Grudt, Study Director — Norwegian University of Science and Technology; Abhijit Sen, prof, Principal Investigator — Norwegian University of Science and Technology; Archana Shrestha, Principal Investigator — Institute for Implementation Sciences and Health, Nepal; Sanju Bhattarai, Principal Investigator — Institute for Implementation Science and Health
Locations (1):
- Institute for Implementation Sciences and Health, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bhattarai S, Shrestha A, Skovlund E, Asvold BO, Mjolstad BP, Sen A. Cluster randomised trial to evaluate comprehensive approach to hypertension management in Nepal: a study protocol. BMJ Open. 2023 May 11;13(5):e069898. doi: 10.1136/bmjopen-2022-069898. PMID 37169495
- [Background] Bhattarai S, Wagle D, Shrestha A, Asvold BO, Skovlund E, Sen A. Role of Perceived Social Support in Adherence to Antihypertensives and Controlled Hypertension: Findings of a Community Survey from Urban Nepal. Patient Prefer Adherence. 2024 Mar 26;18:767-777. doi: 10.2147/PPA.S455511. eCollection 2024. PMID 38558834
- [Background] Bhattarai S, Skovlund E, Shrestha A, Mjolstad BP, Asvold BO, Sen A. Impact of a community health worker led intervention for improved blood pressure control in urban Nepal: an open-label cluster randomised controlled trial. Lancet Reg Health Southeast Asia. 2024 Aug 8;29:100461. doi: 10.1016/j.lansea.2024.100461. eCollection 2024 Oct. PMID 39220804
- [Background] Bhattarai S, Bajracharya S, Shrestha A, Skovlund E, Asvold BO, Mjolstad BP, Sen A. Facilitators and barriers to hypertension management in urban Nepal: findings from a qualitative study. Open Heart. 2023 Oct;10(2):e002394. doi: 10.1136/openhrt-2023-002394. PMID 37899127